CLINICAL TRIAL: NCT05710172
Title: Evaluation of Auditory Mirror-therapy for Tinnitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Nils Clas Linnman, Assistant Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000820
Record Dates: First submitted 2023-01-15; First posted 2023-02-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Masking Description: Concealment of treatment allocation is not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auditory Mirror Therapy Device (Experimental): Modified 3M Peltor Tactical 300 Electronic Hearing Protector. The modification consists of connecting the left microphone to the right microphone tab on the circuit board, and vice versa.
  Interventions: Device: Auditory Mirror Therapy
- Sham Headphone Device (Sham Comparator): Non-Modified 3M Peltor Tactical 300 Electronic Hearing Protector
  Interventions: Device: Auditory Mirror Therapy

INTERVENTIONS:
Device: Auditory Mirror Therapy — 21 days, up to 3 hours per day intervention

SUMMARY:
The investigators will evaluate the effects of wearing auditory mirror earmuffs on tinnitus and on audiometry.The auditory mirror earmuffs is a device that re-routes auditory input from the left side of the head to the right ear, and vice verse, thereby flipping the auditory input. This procedure is called Auditory Mirror Therapy (AMT).

DETAILED DESCRIPTION:
The goal of this study is to determine efficacy of a 21 day, 3 hours per day intervention of auditory mirror therapy (AMT) for chronic tinnitus. Hypothesis: AMT, as contrasted to a sham device, will significantly reduce symptom ratings on the Tinnitus Functional Index (TFI) scale. Along with TFI, additional measures will be collected every two days throughout the intervention; Tinnitus Handicap Index, Visual Analogue Scale, Minimum Masking Level (MML) and Residual Inhibition (RI), and Auditory Mirror Therapy Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages 18-80 years old
* Chronic Tinnitus (> 3months)

Exclusion Criteria:

* Use of hearing aids
* No history of significant drug or alcohol use
* No history of debilitating neurological or psychiatric illnesses
* No current or past history of balance-, vertigo- and/or vestibular- symptoms including Ménières disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Tinnitus Functional Index (TFI) | 3 weeks
  25 question inventory that developed to provide a scaling of tinnitus severity, an identification of tinnitus domains with impact on the tinnitus severity, and a responsive measurement of change in tinnitus severity.
  The TFI will be used to determine the efficacy of a 21 day, 3 hours per day, intervention of auditory mirror-therapy (AMT) for chronic tinnitus

SECONDARY OUTCOMES:
Change in Tinnitus Handicap Inventory (THI) | 3 weeks
  a brief and psychometrically robust self-report measure used to quantify the impact of tinnitus on daily living.
Change in Visual Analogue Scale (VAS) | 3 weeks
  Scale from 0 to 100 for tinnitus awareness, loudness and annoyance, on separate VAS.
  VAS loudness and annoyance are valid and effective measurements for capturing reductions in tinnitus severity in patients with chronic tinnitus
Change in Minimum Masking Level (MML) and residual inhibition (RI) | 3 weeks
  MML is defined as the lowest tone intensity level required to cover or mask and individual's tinnitus.
  Correspondingly, the RI is considered the temporary decrease of tinnitus after a prolonged acoustic stimulation.

OTHER OUTCOMES:
Auditory Mirror Therapy Questionnaire | 3 weeks
  developed to qualitatively analyze how AMT is affecting participants' tinnitus throughout the intervention study. here

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Linnman C. Auditory Mirror Therapy for Tinnitus: A Pilot Study. J Am Acad Audiol. 2022 Apr;33(4):220-223. doi: 10.1055/a-1749-9279. Epub 2022 Dec 6. PMID 35079989